CLINICAL TRIAL: NCT03526289
Title: GIP/GLP-1 Co-Activity in Subjects With Overweight and Type 2 Diabetes: Lowering of Food Intake
Acronym: GASOLIN II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Collaborators: Zealand Pharma (Industry)
Responsible Party: Principal Investigator, Natasha Chidekel Bergmann, Medical doctor, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-16031728
Record Dates: First submitted 2017-10-24; First posted 2018-05-16 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Type 2 Diabetes Mellitus; Overweight and Obesity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GIP infusion (Active Comparator): 5 hours of continuously GIP1-42 infusion
  Interventions: Biological: GIP1-42 infusion
- Saline (Placebo Comparator): 5 hours of continuously saline infusion
  Interventions: Other: Saline

INTERVENTIONS:
Biological: GIP1-42 infusion — 5-hour GIP1-42 infusion (time point 0-300 minutes)
  Arms: GIP infusion
Other: Saline — 5-hour infusion of saline (placebo) (time point 0-300 minutes)
  Arms: Saline

SUMMARY:
The primary aim of the study is to evaluate how GIP receptor activation influence food intake and mechanisms regulating food intake in obese individuals with type 2 diabetes that are in steady treatment with metformin and a GLP-1 receptor agonist.

DETAILED DESCRIPTION:
The study is designed as a double blinded cross-over study with two study days: One day of GIP infusion (for 5 hours) and one day with placebo (saline) infusion (for 5 hours). The primary endpoint is difference in food intake between the two study days. Food intake is examined as amount of food eaten during an ad libitum meal.

ELIGIBILITY:
Inclusion criteria:

* Caucasian men
* Age between 18 and 70 years
* Body mass index (BMI) between 25 and 40 kg/m2
* Type 2 diabetes (diagnosed according to the criteria of the World Health Organization) with HbA1c <69 mM (<8.5 %)
* In stable treatment for ≥3 months with metformin ≥1 g and a GLP-1 receptor agonist.
* Informed consent

Exclusion criteria

* Anaemia (haemoglobin outside normal range)
* Any current or prior gastrointestinal disease that may interfere with the endpoint variables
* Liver disease (alanine aminotransferase (ALAT) and/or serum aspartate aminotransferase (ASAT) > 2 times normal values) or history of hepatobiliary disorder.
* Nephropathy (serum creatinine above normal range and/or albuminuria).
* Anorexia, bulimia or binge eating disorder
* Allergy or intolerance to ingredients included in the standardised meals
* Tobacco smoking
* Treatment with other glucose lowering drugs than GLP-1 receptor agonists and metformin.
* Any regular drug treatment (besides metformin and GLP-1 receptor agonists) that cannot be discontinued for a minimum of 12 hours
* Any physical or psychological condition that the investigator feels would interfere with trial participation

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male fænotype
Enrollment: 22 (Actual)
Dates: Start 2017-11-08 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
food intake | time point 300-330 minutes
  food intake (kJ) eaten from an ad libitum meal of pasta bolognese

SECONDARY OUTCOMES:
Appetite | time point -30, 0, 30, 60, 90, 120, 150, 180, 210, 240, 270 minutes
  Appetite rated on visual analogue scales (0-10 mm)
satiety | time point -30, 0, 30, 60, 90, 120, 150, 180, 210, 240, 270 minutes
  Satiety rated on visual analogue scales (0-10 mm)
prospective food consumption | time point -30, 0, 30, 60, 90, 120, 150, 180, 210, 240, 270 minutes
  prospective food consumption rated on visual analogue scales (0-10 mm)
fullness | time point -30, 0, 30, 60, 90, 120, 150, 180, 210, 240, 270 minutes
  fullness rated on visual analogue scales (0-10 mm)
Thirst | time point -30, 0, 30, 60, 90, 120, 150, 180, 210, 240, 270 minutes
  Thirst rated on visual analogue scales (0-10 mm)
Nausea | time point -30, 0, 30, 60, 90, 120, 150, 180, 210, 240, 270 minutes
  Nausea rated on visual analogue scales (0-10 mm)
Energy expenditure | measured at baseline and at time point 250 minutes
  resting energy expenditure measured by indirect calorimetry (kcal/day)
gastric emptying | ingested at time point -15, 0, 60, 75, 90, 105, 120, 150, 180, 210 and 270 minutes
  acetaminophen test
gallbladder emptying | at time point -15, 0, 30, 60, 90, 120, 150, 180, 240 minutes
  gallbladder emptying evaluated by ultrasound
glucagon responses | at time point -15, 0, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 and 270 minutes
  blood samples
Insulin responses | at time point -15, 0, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 and 270 minutes
  blood samples
C-peptide responses | at time point -15, 0, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 and 270 minutes
  blood samples
gut hormone responses | at time point -15, 0, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 and 270 minutes
  Blood samples
bone turnover markers | at time point -15, 0, 30, 45, 60, 75, 90, 105, 120, 150, 180, 210 and 270 minutes
  Blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Center for diabetes research, Hellerup, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bergmann NC, Gasbjerg LS, Heimburger SM, Krogh LSL, Dela F, Hartmann B, Holst JJ, Jessen L, Christensen MB, Vilsboll T, Lund A, Knop FK. No Acute Effects of Exogenous Glucose-Dependent Insulinotropic Polypeptide on Energy Intake, Appetite, or Energy Expenditure When Added to Treatment With a Long-Acting Glucagon-Like Peptide 1 Receptor Agonist in Men With Type 2 Diabetes. Diabetes Care. 2020 Mar;43(3):588-596. doi: 10.2337/dc19-0578. Epub 2020 Jan 16. PMID 31949084